CLINICAL TRIAL: NCT01404052
Title: Effects of Transcranial Direct Current Stimulation and Transcranial Ultrasound on the Perception of Pain Due to Osteoarthritis of the Knee
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Transcranial Ultrasound on Osteoarthritis Pain of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-p-001977
Record Dates: First submitted 2011-06-29; First posted 2011-07-27 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain; Osteoarthritis
Keywords: transcranial direct current stimulation; transcranial ultrasound
MeSH Terms: conditions — Chronic Pain; Osteoarthritis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + transcranial ultrasound (Experimental): Subjects will undergo 20 minutes active tDCS in conjunction with transcranial ultrasound measurements.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS + transcranial ultrasound (Sham Comparator): Subjects will receive sham tDCS in conjunction with transcranial ultrasound measurements.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Subjects will be randomized to undergo either 5 sessions of active tDCS stimulation, or 5 sessions of sham tDCS stimulation. For both active and sham stimulation, we will use electrodes of 35cm^2 and an intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. Active stimulation will last for 20 minutes, while sham stimulation will only last for 30 seconds, mimicking the sensations during active stimulation.
  Other Names: low intensity 1x1 direct current stimulator

SUMMARY:
The purpose of this study is to see the effects of transcranial direct current stimulation (tDCS) on the pain associated with osteoarthritis of the knee. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation. Before, during and after stimulation, the investigators will measure and assess changes intracranial blood flow with transcranial ultrasound.

ELIGIBILITY:
STUDY ELIGIBILITY CRITERIA

Inclusion Criteria:

1. Providing informed consent to participate in the study
2. 18 to 64 years old
3. Having chronic osteoarthritis knee pain in either knee (existing pain for more than 6 months with an average of at least 3 on a 0-10 VAS scale)
4. Pain resistant to common analgesics and medications for chronic pain such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, and Codeine.
5. Must have the ability to feel pain as self reported

Exclusion Criteria:

1. Subject is pregnant.
2. Contraindications to tDCS:

   * metal in the head
   * implanted brain medical devices
3. Contraindications to TUS:

   * metal in the head
   * implanted brain medical devices
4. History of alcohol or drug abuse within the past 6 months as self reported
5. Use of carbamazepine within the past 6 months as self reported.
6. Suffering from severe depression (with a score of >30 in the Beck Depression Inventory)
7. History of neurological disorders as self reported.
8. History of unexplained fainting spells as self reported,
9. History of head injury resulting in more than a momentary loss of consciousness as self reported
10. History of neurosurgery as self reported

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07-30 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in pain scale | Measured for approximately 2 months
  Determine whether anodal transcranial direct current stimulation in conjunction with transcranial ultrasound (applied in a diagnostic mode) is effective in reducing pain in subjects with chronic osteoarthritis pain, as measured by changes in the Visual Analogue Scale (VAS) for pain. VAS will be measured immediately before the tDCS stimulation sessions, and immediately after the tDCS stimulation sessions for the subject's duration in the trial. VAS will also be measured at baseline, and at three follow-up sessions after tDCS stimulation (up to 2 months after tDCS stimulation)

SECONDARY OUTCOMES:
Changes in cutaneous allodynia/hyperalgesia | Measured for approximately 2 months
  To investigate whether stimulation with active anodal tDCS with ultrasound (applied in a diagnostic mode) alters the phenomenon of central sensitization, as indexed by cutaneous allodynia and hyperalgesia, measured by the pain perception threshold as compared with sham tDCS. Pain measurements will be measured immediately before the tDCS stimulation sessions, and immediately after for the subject's duration in the trial. Pain measurements will also be measured at baseline, and at three follow-up sessions after tDCS stimulation (up to 2 months after tDCS stimulation)
Assessment of hemodynamic changes with transcranial ultrasound | Measured for approximately 2 months
  To investigate hemodynamic changes in the brain that may occur due to tDCS as measured by transcranial ultrasound. Blood flow measured by TUS will be measured immediately before during and after the tDCS stimulation sessions, for the subject's duration in the trial. Blood flow measured by TUS will also be measured at baseline, and at three follow-up sessions after tDCS stimulation (up to 2 months after tDCS stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital (SRH)
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States